CLINICAL TRIAL: NCT04542213
Title: Effect of the Combination of Dipeptidyl Peptidase-4 Inhibitor (DPP4i) and Insulin in Comparison to Insulin on Metabolic Control and Prognosis in Hospitalized Patients With COVID-19
Brief Title: Dipeptidyl Peptidase-4 Inhibitor (DPP4i) for the Control of Hyperglycemia in Patients With COVID-19
Acronym: Covid19DPP4i
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Rodolfo Guardado Mendoza, Principal Investigator, Hospital Regional de Alta Especialidad del Bajio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI-22-2020
Record Dates: First submitted 2020-09-03; First posted 2020-09-09 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Hyperglycemia; Covid19
MeSH Terms: conditions — Hyperglycemia; COVID-19 | interventions — Linagliptin; Insulin

STUDY DESIGN:
Intervention Model Description: The study will include two parallel groups of intervention
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Physicians who will be providing health support will not be aware of the treatment that patients will be receiving regarding this protocol, also the principal investigator and the personal who will be measuring glucose levels and prognosis, will not be aware of the group of treatment, since all the patients will be receiving the same protocol of insulin administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPP4 inhibitor + insulin (Experimental): Patients assigned to this group of treatment will receive Linagliptin 5mg orally once daily plus a basal-bolo insulin scheme
  Interventions: Drug: Linagliptin tablet
- Insulin scheme alone (Active Comparator): Patients assigned to this group will receive only a basal-bolus insulin scheme
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Linagliptin tablet — Linagliptin 5mg once daily plus a basal-bolus insulin scheme
  Other Names: Linagliptin
  Arms: DPP4 inhibitor + insulin
Drug: Insulin — Basal-bolus insulin scheme
  Other Names: Insulin group
  Arms: Insulin scheme alone

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection has been a world health issue during the last months, affecting mostly countries with a high metabolic risk, like Mexico. Patients with type 2 diabetes (T2D) have an increased risk of any kind of infection as well as an increased mortality risk. Hyperglycemia has been established as an important predictor of mortality in patients with T2D and SARS-CoV-2. The standard treatment of hyperglycemia in hospitalized patients has been basen on insulin schemes, but recently evidence suggest the utility of some other drugs, reducing the risk of hypoglucemia and increasing the probability of a proper metabolic control. The goal of this study is to compare the utility of dipeptidyl peptidase-4 inhibitor (DPP4i) as a combination with insulin on metabolic control and prognosis in hospitalized patients with SARS-CoV-2 and hyperglycemia.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection has been a world health issue during the last months, affecting mostly countries with a high metabolic risk, like Mexico. Patients with type 2 diabetes (T2D) have an increased risk of any kind of infection as well as an increased mortality risk. Hyperglycemia has been established as an important predictor of mortality in patients with T2D and SARS-CoV-2. The standard treatment of hyperglycemia in hospitalized patients has been basen on insulin schemes, but recently evidence suggest the utility of some other drugs, reducing the risk of hypoglucemia and increasing the probability of a proper metabolic control. DPP4 enzyme has an ubiquitous distribution and has been considered as a pro-inflammatory enzyme, considering that DPP4 inhibitors could have and anti-inflammatory effect, as it has been shown in different works. The goal os this study is to compare the utility of DPP4 inhibitor as a combination with insulin on metabolic control and prognosis in hospitalized patients with SARS-CoV-2 and hyperglycemia. For this purpose we will randomize patients with SARS-CoV-2 and hyperglycemia to receive either the combination of DPP4i + insulin or insulin alone and will follow al algorithm treatment to define metabolic control as well as prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with confirmed infection by SARS-CoV-2
* Hyperglycemia higher than 140 mg/dl
* Patients accepting oral medications
* Both sex
* Older than 18 years of age
* Patients who accept to participate in the study and sign the consent form

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy
* Hyperosmolar hyperglycemic state or diabetic ketoacidosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Glucose levels | 5-10 days
  Glucose levels during hospitalization
Number of patients who achieve metabolic control | 5-10 days
  Patients who achieve fasting glucose levels below 140 mg/dl and posprandial levels below 180 mg/dl

SECONDARY OUTCOMES:
Number of patients who die or need mechanical ventilation | 5-10 days
  If the patient requires mechanical ventilation or dies
C reactive protein levels | 5-10 days
  C reactive protein measured at basal and at 5-10 days in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Guardado, PhD, Principal Investigator — Hospital Regional de Alta Especialidad del Bajìo
Locations (1):
- Hospital Regional de Alta Especialidad del Bajìo, Leòn, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Sharing of the data can be done, depending on the requested purposes
Supporting Information: Study Protocol
Time Frame: Data will be available once the main results of the study are published, and in accordance with the journal
Access Criteria: Direct contact with the principal investigator

REFERENCES:
- [Background] DeFronzo RA. Pathogenesis of type 2 diabetes mellitus. Med Clin North Am. 2004 Jul;88(4):787-835, ix. doi: 10.1016/j.mcna.2004.04.013. PMID 15308380
- [Background] Levetan CS, Passaro M, Jablonski K, Kass M, Ratner RE. Unrecognized diabetes among hospitalized patients. Diabetes Care. 1998 Feb;21(2):246-9. doi: 10.2337/diacare.21.2.246. PMID 9539990
- [Background] Umpierrez GE, Isaacs SD, Bazargan N, You X, Thaler LM, Kitabchi AE. Hyperglycemia: an independent marker of in-hospital mortality in patients with undiagnosed diabetes. J Clin Endocrinol Metab. 2002 Mar;87(3):978-82. doi: 10.1210/jcem.87.3.8341. PMID 11889147
- [Background] McAlister FA, Majumdar SR, Blitz S, Rowe BH, Romney J, Marrie TJ. The relation between hyperglycemia and outcomes in 2,471 patients admitted to the hospital with community-acquired pneumonia. Diabetes Care. 2005 Apr;28(4):810-5. doi: 10.2337/diacare.28.4.810. PMID 15793178
- [Background] Kes VB, Solter VV, Supanc V, Demarin V. Impact of hyperglycemia on ischemic stroke mortality in diabetic and non-diabetic patients. Ann Saudi Med. 2007 Sep-Oct;27(5):352-5. doi: 10.5144/0256-4947.2007.352. PMID 17921684
- [Background] Angeli F, Verdecchia P, Karthikeyan G, Mazzotta G, Del Pinto M, Repaci S, Gatteschi C, Gentile G, Cavallini C, Reboldi G. New-onset hyperglycemia and acute coronary syndrome: a systematic overview and meta-analysis. Curr Diabetes Rev. 2010 Mar;6(2):102-10. doi: 10.2174/157339910790909413. PMID 20034367
- [Background] Noordzij PG, Boersma E, Schreiner F, Kertai MD, Feringa HH, Dunkelgrun M, Bax JJ, Klein J, Poldermans D. Increased preoperative glucose levels are associated with perioperative mortality in patients undergoing noncardiac, nonvascular surgery. Eur J Endocrinol. 2007 Jan;156(1):137-42. doi: 10.1530/eje.1.02321. PMID 17218737
- [Background] Pomposelli JJ, Baxter JK 3rd, Babineau TJ, Pomfret EA, Driscoll DF, Forse RA, Bistrian BR. Early postoperative glucose control predicts nosocomial infection rate in diabetic patients. JPEN J Parenter Enteral Nutr. 1998 Mar-Apr;22(2):77-81. doi: 10.1177/014860719802200277. PMID 9527963
- [Background] McDonnell ME, Umpierrez GE. Insulin therapy for the management of hyperglycemia in hospitalized patients. Endocrinol Metab Clin North Am. 2012 Mar;41(1):175-201. doi: 10.1016/j.ecl.2012.01.001. Epub 2012 Feb 17. PMID 22575413
- [Background] Stentz FB, Umpierrez GE, Cuervo R, Kitabchi AE. Proinflammatory cytokines, markers of cardiovascular risks, oxidative stress, and lipid peroxidation in patients with hyperglycemic crises. Diabetes. 2004 Aug;53(8):2079-86. doi: 10.2337/diabetes.53.8.2079. PMID 15277389
- [Background] Corathers SD, Falciglia M. The role of hyperglycemia in acute illness: supporting evidence and its limitations. Nutrition. 2011 Mar;27(3):276-81. doi: 10.1016/j.nut.2010.07.013. Epub 2010 Sep 24. PMID 20869205
- [Background] Feng W, Zong W, Wang F, Ju S. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2): a review. Mol Cancer. 2020 Jun 2;19(1):100. doi: 10.1186/s12943-020-01218-1. PMID 32487159
- [Background] Hamming I, Timens W, Bulthuis ML, Lely AT, Navis G, van Goor H. Tissue distribution of ACE2 protein, the functional receptor for SARS coronavirus. A first step in understanding SARS pathogenesis. J Pathol. 2004 Jun;203(2):631-7. doi: 10.1002/path.1570. PMID 15141377
- [Background] Mossel EC, Wang J, Jeffers S, Edeen KE, Wang S, Cosgrove GP, Funk CJ, Manzer R, Miura TA, Pearson LD, Holmes KV, Mason RJ. SARS-CoV replicates in primary human alveolar type II cell cultures but not in type I-like cells. Virology. 2008 Mar 1;372(1):127-35. doi: 10.1016/j.virol.2007.09.045. Epub 2007 Nov 26. PMID 18022664
- [Background] Gheblawi M, Wang K, Viveiros A, Nguyen Q, Zhong JC, Turner AJ, Raizada MK, Grant MB, Oudit GY. Angiotensin-Converting Enzyme 2: SARS-CoV-2 Receptor and Regulator of the Renin-Angiotensin System: Celebrating the 20th Anniversary of the Discovery of ACE2. Circ Res. 2020 May 8;126(10):1456-1474. doi: 10.1161/CIRCRESAHA.120.317015. Epub 2020 Apr 8. PMID 32264791
- [Background] Allard R, Leclerc P, Tremblay C, Tannenbaum TN. Diabetes and the severity of pandemic influenza A (H1N1) infection. Diabetes Care. 2010 Jul;33(7):1491-3. doi: 10.2337/dc09-2215. PMID 20587722
- [Background] Fadini GP, Morieri ML, Longato E, Avogaro A. Prevalence and impact of diabetes among people infected with SARS-CoV-2. J Endocrinol Invest. 2020 Jun;43(6):867-869. doi: 10.1007/s40618-020-01236-2. Epub 2020 Mar 28. No abstract available. PMID 32222956
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Guan WJ, Liang WH, Zhao Y, Liang HR, Chen ZS, Li YM, Liu XQ, Chen RC, Tang CL, Wang T, Ou CQ, Li L, Chen PY, Sang L, Wang W, Li JF, Li CC, Ou LM, Cheng B, Xiong S, Ni ZY, Xiang J, Hu Y, Liu L, Shan H, Lei CL, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Cheng LL, Ye F, Li SY, Zheng JP, Zhang NF, Zhong NS, He JX; China Medical Treatment Expert Group for COVID-19. Comorbidity and its impact on 1590 patients with COVID-19 in China: a nationwide analysis. Eur Respir J. 2020 May 14;55(5):2000547. doi: 10.1183/13993003.00547-2020. Print 2020 May. PMID 32217650
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Cariou B, Hadjadj S, Wargny M, Pichelin M, Al-Salameh A, Allix I, Amadou C, Arnault G, Baudoux F, Bauduceau B, Borot S, Bourgeon-Ghittori M, Bourron O, Boutoille D, Cazenave-Roblot F, Chaumeil C, Cosson E, Coudol S, Darmon P, Disse E, Ducet-Boiffard A, Gaborit B, Joubert M, Kerlan V, Laviolle B, Marchand L, Meyer L, Potier L, Prevost G, Riveline JP, Robert R, Saulnier PJ, Sultan A, Thebaut JF, Thivolet C, Tramunt B, Vatier C, Roussel R, Gautier JF, Gourdy P; CORONADO investigators. Phenotypic characteristics and prognosis of inpatients with COVID-19 and diabetes: the CORONADO study. Diabetologia. 2020 Aug;63(8):1500-1515. doi: 10.1007/s00125-020-05180-x. Epub 2020 May 29. PMID 32472191
- [Background] Bellido V, Suarez L, Rodriguez MG, Sanchez C, Dieguez M, Riestra M, Casal F, Delgado E, Menendez E, Umpierrez GE. Comparison of Basal-Bolus and Premixed Insulin Regimens in Hospitalized Patients With Type 2 Diabetes. Diabetes Care. 2015 Dec;38(12):2211-6. doi: 10.2337/dc15-0160. Epub 2015 Oct 12. PMID 26459273
- [Background] Pasquel FJ, Umpierrez GE. [Management of hyperglycemia in the hospitalized patient]. Medicina (B Aires). 2010;70(3):275-83. Spanish. PMID 20529780
- [Background] Sokos GG, Nikolaidis LA, Mankad S, Elahi D, Shannon RP. Glucagon-like peptide-1 infusion improves left ventricular ejection fraction and functional status in patients with chronic heart failure. J Card Fail. 2006 Dec;12(9):694-9. doi: 10.1016/j.cardfail.2006.08.211. PMID 17174230
- [Background] Guardado-Mendoza R, Cazares-Sanchez D, Evia-Viscarra ML, Jimenez-Ceja LM, Duran-Perez EG, Aguilar-Garcia A. Linagliptin plus insulin for hyperglycemia immediately after renal transplantation: A comparative study. Diabetes Res Clin Pract. 2019 Oct;156:107864. doi: 10.1016/j.diabres.2019.107864. Epub 2019 Sep 17. PMID 31539565
- [Background] Deane AM, Chapman MJ, Fraser RJ, Burgstad CM, Besanko LK, Horowitz M. The effect of exogenous glucagon-like peptide-1 on the glycaemic response to small intestinal nutrient in the critically ill: a randomised double-blind placebo-controlled cross over study. Crit Care. 2009;13(3):R67. doi: 10.1186/cc7874. Epub 2009 May 13. PMID 19439067
- [Background] Mussig K, Oncu A, Lindauer P, Heininger A, Aebert H, Unertl K, Ziemer G, Haring HU, Holst JJ, Gallwitz B. Effects of intravenous glucagon-like peptide-1 on glucose control and hemodynamics after coronary artery bypass surgery in patients with type 2 diabetes. Am J Cardiol. 2008 Sep 1;102(5):646-7. doi: 10.1016/j.amjcard.2008.06.029. No abstract available. PMID 18721530
- [Background] Chakkera HA, Weil EJ, Castro J, Heilman RL, Reddy KS, Mazur MJ, Hamawi K, Mulligan DC, Moss AA, Mekeel KL, Cosio FG, Cook CB. Hyperglycemia during the immediate period after kidney transplantation. Clin J Am Soc Nephrol. 2009 Apr;4(4):853-9. doi: 10.2215/CJN.05471008. Epub 2009 Apr 1. PMID 19339426
- [Background] Broxmeyer HE, Capitano M, Campbell TB, Hangoc G, Cooper S. Modulation of Hematopoietic Chemokine Effects In Vitro and In Vivo by DPP-4/CD26. Stem Cells Dev. 2016 Apr 15;25(8):575-85. doi: 10.1089/scd.2016.0026. Epub 2016 Mar 30. PMID 26943017
- [Background] Mulvihill EE, Drucker DJ. Pharmacology, physiology, and mechanisms of action of dipeptidyl peptidase-4 inhibitors. Endocr Rev. 2014 Dec;35(6):992-1019. doi: 10.1210/er.2014-1035. Epub 2014 Sep 12. PMID 25216328
- [Background] Defronzo RA. Banting Lecture. From the triumvirate to the ominous octet: a new paradigm for the treatment of type 2 diabetes mellitus. Diabetes. 2009 Apr;58(4):773-95. doi: 10.2337/db09-9028. No abstract available. PMID 19336687
- [Background] Guardado-Mendoza R, Salazar-Lopez SS, Alvarez-Canales M, Farfan-Vazquez D, Martinez-Lopez YE, Jimenez-Ceja LM, Suarez-Perez EL, Angulo-Romero F, Evia-Viscarra ML, Montes de Oca-Loyola ML, Duran-Perez EG, Folli F, Aguilar-Garcia A. The combination of linagliptin, metformin and lifestyle modification to prevent type 2 diabetes (PRELLIM). A randomized clinical trial. Metabolism. 2020 Mar;104:154054. doi: 10.1016/j.metabol.2019.154054. Epub 2019 Dec 28. PMID 31887309
- [Background] Meyerholz DK, Lambertz AM, McCray PB Jr. Dipeptidyl Peptidase 4 Distribution in the Human Respiratory Tract: Implications for the Middle East Respiratory Syndrome. Am J Pathol. 2016 Jan;186(1):78-86. doi: 10.1016/j.ajpath.2015.09.014. Epub 2015 Nov 18. PMID 26597880
- [Background] Ploquin MJ, Casrouge A, Madec Y, Noel N, Jacquelin B, Huot N, Duffy D, Jochems SP, Micci L, Lecuroux C, Boufassa F, Booiman T, Garcia-Tellez T, Ghislain M, Grand RL, Lambotte O, Kootstra N, Meyer L, Goujard C, Paiardini M, Albert ML, Muller-Trutwin M. Systemic DPP4 activity is reduced during primary HIV-1 infection and is associated with intestinal RORC+ CD4+ cell levels: a surrogate marker candidate of HIV-induced intestinal damage. J Int AIDS Soc. 2018 Jul;21(7):e25144. doi: 10.1002/jia2.25144. PMID 29987877
- [Background] Seys LJM, Widagdo W, Verhamme FM, Kleinjan A, Janssens W, Joos GF, Bracke KR, Haagmans BL, Brusselle GG. DPP4, the Middle East Respiratory Syndrome Coronavirus Receptor, is Upregulated in Lungs of Smokers and Chronic Obstructive Pulmonary Disease Patients. Clin Infect Dis. 2018 Jan 6;66(1):45-53. doi: 10.1093/cid/cix741. PMID 29020176
- [Background] Thomas L, Eckhardt M, Langkopf E, Tadayyon M, Himmelsbach F, Mark M. (R)-8-(3-amino-piperidin-1-yl)-7-but-2-ynyl-3-methyl-1-(4-methyl-quinazolin-2-ylmethyl)-3,7-dihydro-purine-2,6-dione (BI 1356), a novel xanthine-based dipeptidyl peptidase 4 inhibitor, has a superior potency and longer duration of action compared with other dipeptidyl peptidase-4 inhibitors. J Pharmacol Exp Ther. 2008 Apr;325(1):175-82. doi: 10.1124/jpet.107.135723. Epub 2008 Jan 25. PMID 18223196
- [Background] He YL, Wang Y, Bullock JM, Deacon CF, Holst JJ, Dunning BE, Ligueros-Saylan M, Foley JE. Pharmacodynamics of vildagliptin in patients with type 2 diabetes during OGTT. J Clin Pharmacol. 2007 May;47(5):633-41. doi: 10.1177/0091270006299137. PMID 17442688
- [Background] Heise T, Graefe-Mody EU, Huttner S, Ring A, Trommeshauser D, Dugi KA. Pharmacokinetics, pharmacodynamics and tolerability of multiple oral doses of linagliptin, a dipeptidyl peptidase-4 inhibitor in male type 2 diabetes patients. Diabetes Obes Metab. 2009 Aug;11(8):786-94. doi: 10.1111/j.1463-1326.2009.01046.x. Epub 2009 May 19. PMID 19476474
- [Background] Bergman AJ, Stevens C, Zhou Y, Yi B, Laethem M, De Smet M, Snyder K, Hilliard D, Tanaka W, Zeng W, Tanen M, Wang AQ, Chen L, Winchell G, Davies MJ, Ramael S, Wagner JA, Herman GA. Pharmacokinetic and pharmacodynamic properties of multiple oral doses of sitagliptin, a dipeptidyl peptidase-IV inhibitor: a double-blind, randomized, placebo-controlled study in healthy male volunteers. Clin Ther. 2006 Jan;28(1):55-72. doi: 10.1016/j.clinthera.2006.01.015. PMID 16490580
- [Background] Kim D, Wang L, Beconi M, Eiermann GJ, Fisher MH, He H, Hickey GJ, Kowalchick JE, Leiting B, Lyons K, Marsilio F, McCann ME, Patel RA, Petrov A, Scapin G, Patel SB, Roy RS, Wu JK, Wyvratt MJ, Zhang BB, Zhu L, Thornberry NA, Weber AE. (2R)-4-oxo-4-[3-(trifluoromethyl)-5,6-dihydro[1,2,4]triazolo[4,3-a]pyrazin-7(8H)-yl]-1-(2,4,5-trifluorophenyl)butan-2-amine: a potent, orally active dipeptidyl peptidase IV inhibitor for the treatment of type 2 diabetes. J Med Chem. 2005 Jan 13;48(1):141-51. doi: 10.1021/jm0493156. PMID 15634008
- [Background] Craddy P, Palin HJ, Johnson KI. Comparative effectiveness of dipeptidylpeptidase-4 inhibitors in type 2 diabetes: a systematic review and mixed treatment comparison. Diabetes Ther. 2014 Jun;5(1):1-41. doi: 10.1007/s13300-014-0061-3. Epub 2014 Mar 25. PMID 24664619
- [Background] Del Prato S, Taskinen MR, Owens DR, von Eynatten M, Emser A, Gong Y, Chiavetta S, Patel S, Woerle HJ. Efficacy and safety of linagliptin in subjects with type 2 diabetes mellitus and poor glycemic control: pooled analysis of data from three placebo-controlled phase III trials. J Diabetes Complications. 2013 May-Jun;27(3):274-9. doi: 10.1016/j.jdiacomp.2012.11.008. Epub 2013 Feb 9. PMID 23403068
- [Background] Karagiannis T, Paschos P, Paletas K, Matthews DR, Tsapas A. Dipeptidyl peptidase-4 inhibitors for treatment of type 2 diabetes mellitus in the clinical setting: systematic review and meta-analysis. BMJ. 2012 Mar 12;344:e1369. doi: 10.1136/bmj.e1369. PMID 22411919
- [Background] O'Brien P, O'Connor BF. Seprase: an overview of an important matrix serine protease. Biochim Biophys Acta. 2008 Sep;1784(9):1130-45. doi: 10.1016/j.bbapap.2008.01.006. Epub 2008 Jan 26. PMID 18262497
- [Background] Deacon CF. Dipeptidyl peptidase-4 inhibitors in the treatment of type 2 diabetes: a comparative review. Diabetes Obes Metab. 2011 Jan;13(1):7-18. doi: 10.1111/j.1463-1326.2010.01306.x. PMID 21114598
- [Background] Gross JL, Rogers J, Polhamus D, Gillespie W, Friedrich C, Gong Y, Monz BU, Patel S, Staab A, Retlich S. A novel model-based meta-analysis to indirectly estimate the comparative efficacy of two medications: an example using DPP-4 inhibitors, sitagliptin and linagliptin, in treatment of type 2 diabetes mellitus. BMJ Open. 2013 Mar 5;3(3):e001844. doi: 10.1136/bmjopen-2012-001844. PMID 23468467
- [Background] Egan AG, Blind E, Dunder K, de Graeff PA, Hummer BT, Bourcier T, Rosebraugh C. Pancreatic safety of incretin-based drugs--FDA and EMA assessment. N Engl J Med. 2014 Feb 27;370(9):794-7. doi: 10.1056/NEJMp1314078. No abstract available. PMID 24571751
- [Background] McGuire DK, Alexander JH, Johansen OE, Perkovic V, Rosenstock J, Cooper ME, Wanner C, Kahn SE, Toto RD, Zinman B, Baanstra D, Pfarr E, Schnaidt S, Meinicke T, George JT, von Eynatten M, Marx N; CARMELINA Investigators. Linagliptin Effects on Heart Failure and Related Outcomes in Individuals With Type 2 Diabetes Mellitus at High Cardiovascular and Renal Risk in CARMELINA. Circulation. 2019 Jan 15;139(3):351-361. doi: 10.1161/CIRCULATIONAHA.118.038352. PMID 30586723
- [Background] Rosenstock J, Perkovic V, Johansen OE, Cooper ME, Kahn SE, Marx N, Alexander JH, Pencina M, Toto RD, Wanner C, Zinman B, Woerle HJ, Baanstra D, Pfarr E, Schnaidt S, Meinicke T, George JT, von Eynatten M, McGuire DK; CARMELINA Investigators. Effect of Linagliptin vs Placebo on Major Cardiovascular Events in Adults With Type 2 Diabetes and High Cardiovascular and Renal Risk: The CARMELINA Randomized Clinical Trial. JAMA. 2019 Jan 1;321(1):69-79. doi: 10.1001/jama.2018.18269. PMID 30418475
- [Background] Raj VS, Mou H, Smits SL, Dekkers DH, Muller MA, Dijkman R, Muth D, Demmers JA, Zaki A, Fouchier RA, Thiel V, Drosten C, Rottier PJ, Osterhaus AD, Bosch BJ, Haagmans BL. Dipeptidyl peptidase 4 is a functional receptor for the emerging human coronavirus-EMC. Nature. 2013 Mar 14;495(7440):251-4. doi: 10.1038/nature12005. PMID 23486063
- [Background] Cockrell AS, Peck KM, Yount BL, Agnihothram SS, Scobey T, Curnes NR, Baric RS, Heise MT. Mouse dipeptidyl peptidase 4 is not a functional receptor for Middle East respiratory syndrome coronavirus infection. J Virol. 2014 May;88(9):5195-9. doi: 10.1128/JVI.03764-13. Epub 2014 Feb 26. PMID 24574399
- [Background] Kleine-Weber H, Schroeder S, Kruger N, Prokscha A, Naim HY, Muller MA, Drosten C, Pohlmann S, Hoffmann M. Polymorphisms in dipeptidyl peptidase 4 reduce host cell entry of Middle East respiratory syndrome coronavirus. Emerg Microbes Infect. 2020 Jan 21;9(1):155-168. doi: 10.1080/22221751.2020.1713705. eCollection 2020. PMID 31964246
- [Background] Li K, Wohlford-Lenane C, Perlman S, Zhao J, Jewell AK, Reznikov LR, Gibson-Corley KN, Meyerholz DK, McCray PB Jr. Middle East Respiratory Syndrome Coronavirus Causes Multiple Organ Damage and Lethal Disease in Mice Transgenic for Human Dipeptidyl Peptidase 4. J Infect Dis. 2016 Mar 1;213(5):712-22. doi: 10.1093/infdis/jiv499. Epub 2015 Oct 20. PMID 26486634
- [Background] Peck KM, Cockrell AS, Yount BL, Scobey T, Baric RS, Heise MT. Glycosylation of mouse DPP4 plays a role in inhibiting Middle East respiratory syndrome coronavirus infection. J Virol. 2015 Apr;89(8):4696-9. doi: 10.1128/JVI.03445-14. Epub 2015 Feb 4. PMID 25653445
- [Background] Vankadari N, Wilce JA. Emerging WuHan (COVID-19) coronavirus: glycan shield and structure prediction of spike glycoprotein and its interaction with human CD26. Emerg Microbes Infect. 2020 Mar 17;9(1):601-604. doi: 10.1080/22221751.2020.1739565. eCollection 2020. PMID 32178593
- [Background] Bassendine MF, Bridge SH, McCaughan GW, Gorrell MD. COVID-19 and comorbidities: A role for dipeptidyl peptidase 4 (DPP4) in disease severity? J Diabetes. 2020 Sep;12(9):649-658. doi: 10.1111/1753-0407.13052. Epub 2020 May 27. PMID 32394639
- [Background] Kawasaki T, Chen W, Htwe YM, Tatsumi K, Dudek SM. DPP4 inhibition by sitagliptin attenuates LPS-induced lung injury in mice. Am J Physiol Lung Cell Mol Physiol. 2018 Nov 1;315(5):L834-L845. doi: 10.1152/ajplung.00031.2018. Epub 2018 Sep 6. PMID 30188745
- [Background] Soare A, Gyorfi HA, Matei AE, Dees C, Rauber S, Wohlfahrt T, Chen CW, Ludolph I, Horch RE, Bauerle T, von Horsten S, Mihai C, Distler O, Ramming A, Schett G, Distler JHW. Dipeptidylpeptidase 4 as a Marker of Activated Fibroblasts and a Potential Target for the Treatment of Fibrosis in Systemic Sclerosis. Arthritis Rheumatol. 2020 Jan;72(1):137-149. doi: 10.1002/art.41058. PMID 31350829
- [Background] Beraldo JI, Benetti A, Borges-Junior FA, Arruda-Junior DF, Martins FL, Jensen L, Dariolli R, Shimizu MH, Seguro AC, Luchi WM, Girardi ACC. Cardioprotection Conferred by Sitagliptin Is Associated with Reduced Cardiac Angiotensin II/Angiotensin-(1-7) Balance in Experimental Chronic Kidney Disease. Int J Mol Sci. 2019 Apr 20;20(8):1940. doi: 10.3390/ijms20081940. PMID 31010001
- [Background] Kagal UA, Angadi NB, Matule SM. Effect of dipeptidyl peptidase 4 inhibitors on acute and subacute models of inflammation in male Wistar rats: An experimental study. Int J Appl Basic Med Res. 2017 Jan-Mar;7(1):26-31. doi: 10.4103/2229-516X.198516. PMID 28251104
- [Background] Fadini GP, Morieri ML, Longato E, Bonora BM, Pinelli S, Selmin E, Voltan G, Falaguasta D, Tresso S, Costantini G, Sparacino G, Di Camillo B, Tramontan L, Cattelan AM, Vianello A, Fioretto P, Vettor R, Avogaro A. Exposure to dipeptidyl-peptidase-4 inhibitors and COVID-19 among people with type 2 diabetes: A case-control study. Diabetes Obes Metab. 2020 Oct;22(10):1946-1950. doi: 10.1111/dom.14097. Epub 2020 Jul 1. PMID 32463179
- [Background] Pasquel FJ, Gianchandani R, Rubin DJ, Dungan KM, Anzola I, Gomez PC, Peng L, Hodish I, Bodnar T, Wesorick D, Balakrishnan V, Osei K, Umpierrez GE. Efficacy of sitagliptin for the hospital management of general medicine and surgery patients with type 2 diabetes (Sita-Hospital): a multicentre, prospective, open-label, non-inferiority randomised trial. Lancet Diabetes Endocrinol. 2017 Feb;5(2):125-133. doi: 10.1016/S2213-8587(16)30402-8. Epub 2016 Dec 8. PMID 27964837
- [Background] Umpierrez GE, Gianchandani R, Smiley D, Jacobs S, Wesorick DH, Newton C, Farrokhi F, Peng L, Reyes D, Lathkar-Pradhan S, Pasquel F. Safety and efficacy of sitagliptin therapy for the inpatient management of general medicine and surgery patients with type 2 diabetes: a pilot, randomized, controlled study. Diabetes Care. 2013 Nov;36(11):3430-5. doi: 10.2337/dc13-0277. Epub 2013 Jul 22. PMID 23877988
- [Derived] Guardado-Mendoza R, Garcia-Magana MA, Martinez-Navarro LJ, Macias-Cervantes HE, Aguilar-Guerrero R, Suarez-Perez EL, Aguilar-Garcia A. Effect of linagliptin plus insulin in comparison to insulin alone on metabolic control and prognosis in hospitalized patients with SARS-CoV-2 infection. Sci Rep. 2022 Jan 11;12(1):536. doi: 10.1038/s41598-021-04511-1. PMID 35017617

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04542213/Prot_SAP_000.pdf